CLINICAL TRIAL: NCT00436293
Title: A Randomized Phase II Study of Concurrent Cisplatin-radiotherapy With or Without Neoadjuvant Chemotherapy Using Taxotere and Cisplatin in Advanced Nasopharyngeal Carcinoma (NPC)
Brief Title: Taxotere + Cisplatin in Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_6002
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin

ARMS (2):
- 1 (Experimental): Neo-adjuvant Taxotere followed by cisplatin and radiotherapy
  Interventions: Drug: Docetaxel
- 2 (Active Comparator): Cisplatin and radiotherapy alone without neo-adjuvant chemotherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m²
  Arms: 1
Drug: Cisplatin — 75 mg/m²
  Arms: 2

SUMMARY:
Primary objective:

To assess and compare the toxicities of patients with advanced NPC treated with concurrent cisplatin-radiotherapy with or without neoadjuvant Taxotere (docetaxel) and cisplatin.

Secondary objective:

To assess tumor control and survival

ELIGIBILITY:
Inclusion Criteria:

* International Union against Cancer stages III and IV newly diagnosed NPC

Exclusion Criteria:

* Inadequate bone marrow reserve
* Inadequate renal function
* Other primary malignancy
* Evidence of distant metastases

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Treatment response is evaluated by correlating findings on clinical examination, endoscopy, biopsy, Computed tomography or Magnetic resonance imaging as appropriate. | From administration of drug to end of study

SECONDARY OUTCOMES:
Adverse Events | From administration of drug to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Hong Kong, Hong Kong